CLINICAL TRIAL: NCT06477133
Title: A Randomized, Controlled Trial of Magnesium Sulfate as an Adjunctive Analgesic in Prostate Surgery
Brief Title: Magnesium Sulfate as an Adjunctive Analgesic in Prostate Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-00463
Record Dates: First submitted 2024-06-20; First posted 2024-06-27 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Prostatectomy
Keywords: Prostate surgery; analgesia
MeSH Terms: conditions — Agnosia | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Magnesium (Experimental): Patients in the first group will receive 2 grams magnesium sulfate at the end of surgery as a bolus over approximately 10 minutes intravenously.
  Interventions: Drug: Magnesium sulfate
- No magnesium (No Intervention): Patients in the second group will receive no magnesium.

INTERVENTIONS:
Drug: Magnesium sulfate — Pre-mixed solution of 2 grams of magnesium sulfate dissolved in 20 mL sterile water
  Arms: Magnesium

SUMMARY:
The purpose of this clinical trial is to determine if receiving magnesium sulfate as an adjunctive analgesic for prostate surgery is effective in reducing pain. Subjects will be randomized to receive magnesium or not receive it, as part of a standardized general anesthetic for prostate surgery. The primary objective is to demonstrate improved pain scores in patients receiving magnesium sulfate as an adjunctive analgesic during surgery. Secondary objectives include demonstrating reduced requirements for other opioids, reduced postoperative shivering, improved discharge home and adequate neuromuscular blockade reversal, measured by quantitative train of four monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older.
2. Undergoing a robotic prostatectomy under general anesthesia.
3. Is willing and able to provide consent to participate in the study.

Exclusion Criteria:

1. Patients younger than 18 years
2. Patients with end-stage renal disease
3. Known allergy to magnesium sulfate preparations
4. Any patient that the investigators feel cannot comply with all study related procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain score | 30 minutes after awakening from anesthesia
  Patients will be asked to assess their pain based on a 10-point scale, where 0=no pain and 10=worst imaginable pain.

SECONDARY OUTCOMES:
Pain score | 60 minutes after awakening from anesthesia
  Patients will be asked to assess their pain based on a 10-point scale, where 0=no pain and 10=worst imaginable pain.
Pain score | 120 minutes after awakening from anesthesia
  Patients will be asked to assess their pain based on a 10-point scale, where 0=no pain and 10=worst imaginable pain.
Number of participants who experienced nausea or vomiting | Up to 120 minutes after awakening from anesthesia
Number of participants who experienced postoperative shivering | Up to 120 minutes after awakening from anesthesia
Number of participants who received analgesics in the post anesthesia care unit (PACU) | Through PACU stay, on average 2 hours
Time to administration of analgesics | From awakening from anesthesia to administration of analgesic, up to 120 minutes postoperative
Dose of opioid analgesia given | Through PACU stay, on average 2 hours
  Dose of opioid analgesia given will be measured in milligram morphine equivalents
Number of patients who were admitted to the hospital | From PACU admission to discharge, up to 120 minutes postoperative
Number of patients who were discharged home | From PACU admission to discharge, up to 120 minutes postoperative
Train-of-four (TOF) ratio | TOF ratios will be measured for the duration of the operation, approximately 3 hours
  Train- of-four ratio (TOF) is the ratio of the fourth muscle response to the first one.

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Nunnally, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research, provided the investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at (Link to be provided). The protocol, Statistical Analysis Plan, and Informed Consent Form will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting requests and accessing data may be found at (Link to be provided).